CLINICAL TRIAL: NCT03151070
Title: Scaling Up an Integrated Approach to Improve Delivery Care and Reduce Maternal and Perinatal Mortality in North Guatemala With Stepped Wedge Design
Brief Title: Scaling Up an Integrated Approach to Improve Delivery Care in North Guatemala With Stepped Wedge Design
Acronym: QVLM
Status: Completed | Type: Observational
Sponsor: Hospital San Juan de Dios Guatemala (Other Government)
Collaborators: Grand Challenges Canada (Other); PRONTO International (Unknown)
Responsible Party: Principal Investigator, Edgar Kestler, Executive Director of Epidemiological Research Center in Sexual and Reproductive Health, Hospital San Juan de Dios Guatemala
Other Study IDs: CIESARQVLM17
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Maternal Sepsis During Labor; Hemorrhage, Postpartum; Eclampsia; Complicating Pregnancy; Pre-Eclampsia; Perinatal Morbidity
MeSH Terms: conditions — Postpartum Hemorrhage; Eclampsia; Pregnancy Complications; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Zone 1: Zone 1 includes the following communities from Huehuentenango Distric:
  * San Rafael Petzal
  * San Sebastian Huehuetenango
  * San Gaspar Ixchil
  * Santa Bárbara
  * Colotenango
  * Aguacatán
  Interventions: Other: QVLM Intervention package
- Zone 2: Zone 2 includes the following communities from Alta Verapaz district:
  * Tamahú
  * San Miguel Tucurú
  * Panzós
  * Senahú
  * Telemán
  Interventions: Other: QVLM Intervention package
- Zone 3: Zone 3 includes the following communities from Huehuetenango district:
  * San Idelfonso Ixtahuacán
  * La Democracia
  * San Juan Atitán
  * Tectitán
  * Santiago Chimaltenango
  Interventions: Other: QVLM Intervention package
- Zona 4: Zone 4 includes the following communities from Alta Verapaz district:
  * Lanquín
  * Santa María Cahabón
  * Chisec
  * Chahal
  * Raxruhá
  * Campur
  Interventions: Other: QVLM Intervention package
- Zona 5: Zone 5 includes the following communities from Huehuetenango district:
  * Nenton
  * Jacaltenango
  * Todos Santos Cuchumatán
  * Santa Eulalia
  * San Mateo Ixtatán
  * San Juan Ixcoy
  Interventions: Other: QVLM Intervention package
- Zona 6: Zone 6 includes the following communities from Alta Verapaz district:
  * Santa Cruz Verapaz
  * Tactic
  * San Pedro Carchá
  * San Juan Chamelco
  Interventions: Other: QVLM Intervention package

INTERVENTIONS:
Other: QVLM Intervention package — QVLM intervention package consists of 3 simultaneous interventions:
  * Social marketing to promote insitutional deliveries.
  * PRONTO training to public health personnel
  * Improve interaction with traditional birth attendants

SUMMARY:
"¡Que Vivan las Madres!: Venga a tener su parto al CAP" (QVLM) is a guatemalan quasi-experimental study that has been performed from January 2014 to January 2017 by the Epidemiological Research Center in Sexual and Reproductive Health (CIESAR) in Guatemala in coordination with PRONTO International and University of San Francisco, California. This project has been financed by Grands Challenges Canada' "Save Lives at Birth, A Grand Challenge for Development" partnership that includes USAID, Norwegian ministry of foreign affairs, Bill&Melinda Gates foundation, UKaid. This project has applied a stepped wedge design (SWD) over 6 zones or clusters. Each one of the zones contains from 4 to 6 communities, each one with the presence of one second level health facility (known in Spanish as CAP, Centro de Atención Permanente). These health centers are the next level in attention after home, traditional and empirical attention. Communities around the selected health centers are mostly rural and have the worst maternal health indicators in the country. These health centers are expected to have enough equipment and personnel to attend the deliveries that occur in their communities. This study was performed in Huehuetenango and Alta Verapaz districts in north Guatemala. Each one with 3 zones for a total of 6 zones. The study follows a Stepped Wedge Design, in which all 6 zones are eventually intervened, but at different regular periods of time (each period is 4 months long). This project applies a package of 3 simultaneous interventions in each zone with the purpose of increasing institutional deliveries and improving deliveries attention in public health centers. This intervention plan has been implemented in a pilot study reported in (Kestler et. al, 2013).

DETAILED DESCRIPTION:
Individual delivery data has been collected in site from health centers records. Thus, the study does not depend on official data from the ministry of health. Not only is MOH data hard to obtain, it also may not contain the details we are interested in that are put by hand by doctors and nurses in clinic histories. In order to get uniform data that fits the study needs, a parallel monitoring process has been set up. Data for mortality and morbidity events that occured in communities during the study is limited. We don't have the community counterpart of our indicators. Government data of perinatal deaths in community may be obtained with 1 or 2 years of delay, however there may be an underreporting of such events. Likewise, there is no data source for maternal morbidity in community deliveries since community practice is usually not documented nor reported.

The concept of perinatal mortality used in this study is not the standard concept that includes death from 28th gestational week to 7 days after birth. The perinatal mortality outcome in this study takes into account only deaths that occur during care in health centers (approximately 48 hours since birth). This is intentional since the aim of this study is to improve clinics' skilled delivery care, thereferore it is concerned on reducing the newborn deaths that occur during care given in site. Along this study, the focus is in these subset of perinatal deaths.

The APGAR measure 1 minute and 5 minutes after birth, and the reported procedures for the newborn are used to identify cases of perinatal morbidity.

This study is targetted to the low level health centers in Huehuetenango and Alta Verapaz. This includes 33 health centers. This is a fixed number of health centers and there is no control of the patients that got treated at the health centers. This is the reason why there is no sample size assessment. The selection of the health centers was limited by the definition of CAP (second level health facilities according to local definition) and the amount of patients that received the intervention by attending their deliveries in health centers can not be controlled.

Having data on all vaginal and uncomplicated deliveries that occur in health centers, the analysis can be done by individual cases and also by aggregating data in time periods. Also, analysis methodology of trials with stepped wedge design has been developed in the last years. A generalized mixed model for a multilevel and longitudinal analysis is going to be used in order to account for different sources of variability within and between health centers and times. So far (April 2017) we have done preliminary analysis this way and are confortable with this methodology selection.

ELIGIBILITY:
Inclusion Criteria:

* For participating facilities, health centers in Huehuetenango and Alta Verapaz districts.
* For participating facilities, health centers of type "CAP" (centro de atención permanente) which is the second level of attention in Guatemala, after attention in home and community.
* For institutional deliveries events, vaginal deliveries attended in participating health centers.
* For perinatal morbidity and mortality, any child that is born from an eligible vaginal delivery.

Exclusion Criteria:

* For deliveries, cesarean sections are ignored, since the training is focused on vaginal delivery care.
* In a secondary analysis, perinatal mortality cases that occured before arrival to the health center are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The total population projected for 2014 for the involved communities is approximately 1.4 million. Each community is associated to one low level public health center. Communities in Huehuetenango have an average population of 34,158, and those in Alta Verapaz have 61,237. In the 33 communities, 75% of live births occurred at home while only 22% of live births had medical attention according to national live birth data from 2014. Huehuetenango district has perinatal mortality rate of 43 (per 100,000 live births) and Alta Verapaz district has 35. These two districts have the worst perinatal mortality indicators according to the guatemalan national survey on maternal and child health (ENSMI) for the period 2014-2015.
Sampling Method: Non-Probability Sample
Enrollment: 32000 (Actual)
Dates: Start 2013-12-15 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Mother morbidity | January 2014 - January 2017
  Presence of any of the following conditions: post-partum hemorrhage, eclampsia, pre-eclampsia and sepsis.
Perinatal morbidity | January 2014 - January 2017
  APGAR 1 and 5 minutes after birth. Special attention after birth (resucitation, AMBU and cardiac massage)
Perinatal mortality | January 2014 - January 2017
  Death of the newborn during attention in the health center.
Counts of institutional deliveries | January 2014 - January 2017
  Monthly counts of institutional deliveries in each health center.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Kestler, Msc, Study Director — Researh Center Director

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kestler E, Walker D, Bonvecchio A, de Tejada SS, Donner A. A matched pair cluster randomized implementation trail to measure the effectiveness of an intervention package aiming to decrease perinatal mortality and increase institution-based obstetric care among indigenous women in Guatemala: study protocol. BMC Pregnancy Childbirth. 2013 Mar 21;13:73. doi: 10.1186/1471-2393-13-73. PMID 23517050
- [Background] Walker DM, Holme F, Zelek ST, Olvera-Garcia M, Montoya-Rodriguez A, Fritz J, Fahey J, Lamadrid-Figueroa H, Cohen S, Kestler E. A process evaluation of PRONTO simulation training for obstetric and neonatal emergency response teams in Guatemala. BMC Med Educ. 2015 Jul 24;15:117. doi: 10.1186/s12909-015-0401-7. PMID 26206373
- [Background] Hemming K, Lilford R, Girling AJ. Stepped-wedge cluster randomised controlled trials: a generic framework including parallel and multiple-level designs. Stat Med. 2015 Jan 30;34(2):181-96. doi: 10.1002/sim.6325. Epub 2014 Oct 24. PMID 25346484